CLINICAL TRIAL: NCT04708080
Title: Effect of Thoracic Epidural Analgesia on Short-term Outcome and Mortality in Geriatric Patients With Open Heart Surgery
Brief Title: Effects of Thoracic Epidural Analgesia in Geriatric Patients Undergoing Open Heart Surgery
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ali AKDOĞAN, assistant professor, Karadeniz Technical University
Other Study IDs: 2020/182
Record Dates: First submitted 2021-01-08; First posted 2021-01-13 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Epidural Analgesia; Mechanical Ventilation; Postoperative Complications; Analgesia
Keywords: thoracic epidural analgesia; Postoperative Complications; mortality; Mechanical Ventilation; open heart surgery
MeSH Terms: conditions — Postoperative Complications; Agnosia | interventions — Tea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group E: patients who underwent thoracic epidural catheter for postoperative analgesia
  Interventions: Procedure: thoracic epidural analgesia
- Group I: Patients who cannot be applied thoracic epidural catheter for postoperative analgesia

INTERVENTIONS:
Procedure: thoracic epidural analgesia — A thoracic epidural catheter is routinely placed in patients undergoing open heart surgery in our hospital, at least 1 hour before heparin administration during the operation. After standard monitoring (ECG, SpO2, NIBP) is applied to the patients in the operating room, sedoanalgesia is provided with 1-3mg of midazolam and 50-100mcg of fentanyl. Then, by providing sterilization conditions, an epidural catheter is inserted through the T5-T6 interval with Tuohy needle. After confirming the location of the epidural catheter, 25mg / 10ml bupivacaine is administered as a bolus and then 3ml / hour bupivacaine infusion is started from the solution prepared as 3mg / ml and continues until the 48th postoperative hour. On the postoperative 2nd day, the catheter is removed 10-12 hours after LMWH administration and 2-4 hours after UFH, as recommended by the guidelines, paying attention to the anticoagulant administration times applied to the patients.
  Groups: Group E

SUMMARY:
Elderly patients have a higher incidence of morbidity and mortality due to the interaction of various factors such as decreased physiological reserves, concomitant comorbidities, multiple drug use, cognitive dysfunction, and frailty. Surgical stress, pain and associated lung complications are common problems in open heart surgeries that can affect morbidity and mortality. With a good postoperative pain control and improved respiratory mechanics, complications that may develop in patients can be significantly prevented, and the hospital cost can be reduced and the workforce loss of patients can be reduced by reducing the length of hospital stay in the intensive care unit. Thoracic epidural analgesia (TEA) is an anesthetic analgesia method that has positive effects on many organ systems as well as providing good pain control and is frequently used in open heart surgery. The aim of this study is to investigate the effects of TEA on postoperative respiratory mechanics in geriatric patients, based on analgesia levels, extubation times, length of stay in intensive care, arterial blood gases, morbidity and mortality.

DETAILED DESCRIPTION:
It has been shown that stress response suppression by providing good analgesia with local or systemic methods in the postoperative period reduces mortality and morbidity in many types of surgery. Especially the physiological changes that occur with aging, comorbid diseases and the drugs used in the treatment of these diseases, the type of surgery performed, the postoperative pain treatment and the anesthesia method chosen affect mortality and morbidity Thoracic epidural analgesia (TEA) has provided similar benefits in open heart surgery by suppressing stress response and increasing functional residual capacity with positive effects on the diaphragm, as well as providing good analgesia with thoracic sympathetic block.TEA has positive effects on postoperative pulmonary and circulatory system in selected eligible patients; It allows earlier extubation and provides excellent analgesia. It has been reported that TEA combined with general anesthesia in elective cardiac surgery offers a significant advantage compared to general anesthesia in terms of intensive care and hospital stay, improvement or morbidity. Studies have shown that TEA reduces surgical stress response, improves hemodynamic stability, and reduces the incidence of myocardial ischemia after coronary artery bypass surgery (CABG) as well as supraventricular arrhythmias in the postoperative period .

Based on these studies, the investigators determined the effects of TEA combined with general anesthesia on postoperative respiratory mechanics, analgesia levels, extubation times, length of stay in intensive care, arterial blood gases, effects on organ functions, morbidity and mortality in geriatric patients with open heart surgery in our hospital. the investigators aimed to contribute to the literature by reviewing it retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Elective patients undergoing open heart surgery

Exclusion Criteria:

* Emergency operations
* Patients whose data cannot be reached
* Patients younger than 65
* Patients whose records could not be accessed and who were excluded from the study group procedure in which they were included for any reason will not be included in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study was planned as a retrospective (retrospective) study involving patients aged 65 and over who underwent elective open heart surgery between January 1, 2008 and December 31, 2019.
Sampling Method: Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
the effect of thoracic epidural analgesia | up to 4 weeks
  postoperative respiratory parameters
the effect of thoracic epidural analgesia | postoperative period 3 day
  Patients' sedation and analgesia levels
the effect of thoracic epidural analgesia | 1 day
  extubation times
the effect of thoracic epidural analgesia | 1 month
  postoperative respiratory complications
the effect of thoracic epidural analgesia | up to 4 weeks
  lengths of ICU and hospitality stay
the effect of thoracic epidural analgesia | 1 year
  mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)